CLINICAL TRIAL: NCT03986437
Title: A Prospective Study to Collect Images in Patients Treated With Iodine-131 as Part of a European Research Project in Radiation Protection.
Acronym: MEDIRAD
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 19VADS05
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2020-05

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Differentiated Thyroid Cancer; Iodine-131; Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial is a prospective, non-interventional, monocentric study aiming to collect standard of care imaging of patients treated with Iodine-131 for the determination of dosimetric studies.

Data from this study will be collected as part of an European research project called MEDIRAD.

The overall objectives of this project are to enhance the scientific bases and clinical practice of radiation protection in the medical field, and more specifically to develop and implement the tools necessary to establish the range of absorbed doses delivered to healthy organs in patients undergoing thyroid ablation and the threshold absorbed dose required for thyroid ablation. This will enable patient specific treatment planning that will minimize risk to the patient while ensuring a successful outcome and will facilitate development of a large scale epidemiological study of the effect of low absorbed doses from irradiation of normal organs with internal sources of radionuclides.

Patients will be followed as part of their standard of care. Imaging (SPECT/CT (Single Photon Emission Computed Tomography-Computerized Tomography) and Whole Body scintigraphy) performed at 48 hours post Iodine-131 treatment will be collected. Measures of external gamma radiation will also be collected in the European database.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with differentiated thyroid cancer (papillary or follicular) stage T1b, T2, T3A, Nx-N0-N1, M0 (according to AJCC 8th edition, 2017) of intermediate risk of recurrence (according to 2015 ATA Risk Stratification System)
2. Patient is eligible to receive a therapeutic activity of 3.7 GBq of I-131 after total thyroidectomy or completion thyroidectomy
3. Age ≥ 18 years old
4. Patient affiliated to the French social security system
5. Patient who has received an informed consent for the study

Exclusion Criteria:

1. Patient who has received an external radiotherapy within 6 weeks prior to I-131 treatment
2. Patient who has received a systemic chemotherapy within 6 weeks prior to I-131 treatment
3. History of treatment with I-131
4. Pregnant or breastfeeding women
5. Any psychological, familial, geographical or sociological condition potentially preventing the medical follow-up and/or study procedures
6. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with differentiated thyroid cancer and who are eligible for a Iodine-131 (I-131) treatment after a total thyroidectomy or completion thyroidectomy will be invited to join the study.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with interpretable images | 1 week per patient

SECONDARY OUTCOMES:
Rate of radiation dose | 1 week per patient

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France